CLINICAL TRIAL: NCT03622671
Title: Association of Fibrin Clot Properties With Blood Loss Following Coronary Artery By-pass Grafting - Does Surgical Technique of Left Internal Mammary Artery Harvesting Matter
Brief Title: Fibrin Clot Properties and Blood Loss Following Coronary Artery By-pass Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Piotr Mazur, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: K/ZDS/007961
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease; Internal Mammary-Coronary Artery Anastomosis; Coronary Artery Bypass; Blood Loss, Postoperative; Fibrinolysis
Keywords: Coronary Artery By-pass Grafting; CABG; Fibrin; Clot Lysis Time; CLT; Bleeding; Drainage; Rethoracotomy
MeSH Terms: conditions — Coronary Artery Disease; Postoperative Hemorrhage; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with parallel group design. Equal allocation.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded to LIMA harvesting technique. The laboratory technicians will be blinded to LIMA harvesting technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skeletonized LIMA (Active Comparator): In patients in this arm the left internal mammary artery will be skeletonized without opening of the left pleural cavity during CABG.
  Interventions: Procedure: Skeletonized LIMA
- Pedicled LIMA (Active Comparator): In patients in this arm the left internal mammary artery will be harvested as a pedicled graft with wide opening of left pleural cavity.
  Interventions: Procedure: Pedicled LIMA

INTERVENTIONS:
Procedure: Skeletonized LIMA — Standard CABG - no different form any other procedure of this type except LIMA will be skeletonized without opening the pleura
  Arms: Skeletonized LIMA
Procedure: Pedicled LIMA — Standard CABG - no different form any other procedure of this type except LIMA will be taken down as a pedicled graft with opening the pleura
  Arms: Pedicled LIMA

SUMMARY:
Up to 15% of operations in cardio-pulmonary by-pass are complicated by excessive postoperative blood loss, which negatively affects the outcomes. Recently, it has been demonstrated that fibrin clot susceptibility to lysis is a modulator of postoperative blood loss after cardiac surgery for aortic stenosis. Earlier, a preliminary study showed a negative association of postoperative blood loss after coronary artery by-pass grafting (CABG) with fibrin clot lysis time, reflecting susceptibility to fibrinolysis.

In CABG, postoperative blood loss may depend on the operative technique with respect to left internal mammary artery (LIMA) harvesting. LIMA is taken down in virtually all CABG procedures, but harvesting technical details remain at surgeons discretion (skeletonization without opening the pleural cavity vs. pedicled graft with pleura wide open).

The investigators decided to test the hypothesis that fibrin clot properties modulate the postoperative drainage following CABG strongly enough to attenuate the influence of surgical technique by randomizing the patients undergoing CABG with regard to LIMA harvesting technique.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically confirmed coronary artery disease
* Heart Team qualification for first time elective coronary artery by-pass grafting
* No significant valvular disease or congenital heart disease
* Normal sinus rhythm on ECG
* Continued aspirin in perioperative period

Exclusion Criteria:

* Need for any concomitant cardiac procedure
* St. p. percutaneous coronary intervention within preceding 3 months
* Any previous cardiac surgery
* Known bleeding diathesis
* Acute cardiovascular incident within preceding 3 months
* Heart failure with left ventricular ejection fraction <30%
* Any autoimmune disease
* Any acute infection
* Known neoplasm
* Any thyroid disease
* Treatment with any thienopyridine, oral anticoagulant, heparin or any non-steroid anti-inflammatory agent other than aspirin
* Mental disorder
* Severe comorbidities (liver failure, renal failure on hemodialysis)
* Lacking consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Postoperative chest-tube output after 12 hours | 12 hours from the end of operation
  Drainage volume after 12 hours

SECONDARY OUTCOMES:
Perioperative myocardial infarction | 48 hours after the procedure
  Change in myocardial necrosis biomarkers (Troponin T, creatine kinase) during first 48 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Mazur, MD, Principal Investigator — Jagiellonian University
Locations (1):
- The John Paul II Hospital, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided